CLINICAL TRIAL: NCT04233957
Title: The Role of Oxidative Stress and Endothelial Dysfunction in High Sodium-Induced Changes in Pulsatile Hemodynamics
Brief Title: Dietary Sodium, Oxidative Stress, and Pulsatile Hemodynamics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1452626
Record Dates: First submitted 2019-12-23; First posted 2020-01-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sodium Excess
Keywords: endothelium; oxidative stress; physical activity; ventricular-vascular coupling; pulsatile load
MeSH Terms: conditions — Hypernatremia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Sodium (Experimental): Consumption of an extra 3900 mg of dietary sodium per day.
  Interventions: Dietary Supplement: High Sodium
- Placebo (Placebo Comparator): Control Condition
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: High Sodium — 10 days of 3900 mg of sodium/day in excess of normal dietary intake delivered via enteric capsules filled with table salt.
  Arms: High Sodium
Other: Placebo — 10 days of enteric capsules filled with dextrose.
  Arms: Placebo

SUMMARY:
High sodium diets impair vascular function, which may influence the work of the heart. This investigation is designed to determine if this change in vascular function results in a greater workload in the heart and if people who regularly exercise are protected from these effects.

DETAILED DESCRIPTION:
Excess dietary sodium is associated with cardiac hypertrophy independent of changes in blood pressure. Importantly, increased arterial pulsatile load predicts left ventricular hypertrophy, and thus presents a potential mechanism through which high dietary sodium augments cardiovascular disease risk.

While high sodium diets impair vascular function via an increase in oxidative stress, how high sodium influences central pulsatile hemodynamics is not known. This project aims to a) determine how impaired vascular function affects pulsatile hemodynamics and thus influences the work of the heart during periods of high sodium consumption and b) examine whether regular aerobic exercise and/or fitness protects against the deleterious effects of excess sodium.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (age 21-45) who are either sedentary (1 or less days of exercise per week during past year) or habitually active (4 or more days of aerobic exercise per week for a minimum of 1 year)

Exclusion Criteria:

* Body mass index <18 or >35
* Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90
* Blood donation within past 8 weeks,
* Glucose 6 phosphate dehydrogenase (G6PD) deficiency
* A history of cancer, diabetes, or any other chronic disease
* A history of any heart disease
* A history of hormone therapy
* Use of nicotine products
* Pregnancy
* Nursing mothers
* Participation in regular physical activity greater than 1 day/week- but less than 4 days/week

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reflected Pulse Wave Amplitude | On the 10th day of each arm.
  Aortic pressure-flow relations will be assessed non-invasively using echocardiography and peripheral artery applanation tonometry. Wave separation analysis will be used to calculate reflected pulse wave amplitude.
Conduit artery endothelium-dependent dilation | On the 10th day of each arm.
  Brachial artery flow mediated dilation (FMD) will be assessed by duplex ultrasound as an index of conduit artery endothelial function.
Arterial Stiffness | On the 10th day of each arm.
  Carotid-femoral pulse wave velocity (cf-PWV) will be assessed via applanation tonometry as an index of aortic stiffness. cf-PWV will be calculated as the difference in timing of of pulse waves at the carotid and femoral arteries divided by the distance between measurements.

SECONDARY OUTCOMES:
Wave reflection timing | On the 10th day of each arm.
  Aortic pressure-flow relations will be assessed non-invasively using echocardiography and peripheral artery applanation tonometry. Wave separation analysis will be used to calculate reflected wave transit time.
Forward Pulse Wave Amplitude | On the 10th day of each arm.
  Aortic pressure-flow relations will be assessed non-invasively using echocardiography and peripheral artery applanation tonometry. Wave separation analysis will be used to the amplitude of the forward traveling pulse wave.
24 Hour Blood Pressure | The morning of day 9 through the morning of day 10 for each arm.
  24 hour blood pressure monitoring will be performed using an ambulatory blood pressure monitor device. Average day and nighttime systolic, diastolic, and mean blood pressures will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: David G Edwards, PhD, Principal Investigator — University of Delaware
Locations (1):
- Department of Kinesiology and Applied Physiology, University of Delaware, Newark, Delaware, United States